CLINICAL TRIAL: NCT05991947
Title: Preliminary Experimental Study on Key Technologies for Early Screening of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Secretary of the party committee, Zhejiang Cancer Hospital
Other Study IDs: IRB-2023-427
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer; Healthy
Keywords: Gastric Cancer; Proteomics; Diagnostic model
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- gastric cancer patients
  Interventions: Other: No intervention
- healthy individuals
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention measures are needed.

SUMMARY:
This project aims to collect peripheral blood samples from newly diagnosed gastric cancer patients and healthy individuals. Various techniques such as cfDNA sequencing, proteomics, and fragmentomics will be employed to analyze differences in the expression of ctDNA mutations, fragmentomics, and protein biomarkers between gastric cancer patients and healthy individuals. A new comprehensive diagnostic model will be established and its diagnostic value (sensitivity, specificity, accuracy, etc.) for gastric cancer will be validated.

Specifically, the study will involve the following subjects and quantities: 700 participants from Zhejiang Cancer Hospital (350 gastric cancer patients and 350 healthy individuals), 200 participants from Sichuan Cancer Hospital (100 gastric cancer patients and 100 healthy individuals), and 200 participants from the Sixth Affiliated Hospital of Sun Yat-sen University (100 gastric cancer patients and 100 healthy individuals). Peripheral blood samples (a total of 15mL from each participant, collected in 3 tubes) will be collected from all subjects. The collected blood samples will undergo multi-omics sequencing including cfDNA methylation sequencing, proteomics, and genomics to establish a multi-omics-based early diagnostic model.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 100 years.
* ECOG performance status of 0 or 1.
* Pathologically confirmed Stage I-III gastric cancer patients.
* Patients who have not undergone any anti-tumor treatment (including chemotherapy, radiotherapy, targeted therapy, surgery, anesthesia, etc.) before blood collection.
* Subjects and their family members who can comprehend the research protocol and are willing to participate in the study, providing written informed consent.

Exclusion Criteria:

* Presence of other hereditary diseases or other tumors.
* Severe inflammatory reactions caused by acute illnesses within 14 days prior to blood draw or use of steroids.
* Previous organ transplantation, stem cell transplantation, bone marrow transplantation, or blood transfusion within the last month before enrollment.
* Pregnant women.
* Participation in other clinical trials requiring medication intake within the last 60 days (including anesthesia).
* Severe cardiovascular diseases, uncontrolled infections, or other uncontrollable comorbidities.
* Subjects or family members unable to comprehend the conditions and objectives of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Number of Participants and Total Enrollment:
  Zhejiang Cancer Hospital: 700/700 (350 cases of gastric cancer patients, 350 cases of healthy individuals) Sichuan Cancer Hospital: 200/200 (100 cases of gastric cancer patients, 100 cases of healthy individuals) The Sixth Affiliated Hospital of Sun Yat-sen University: 200/200 (100 cases of gastric cancer patients, 100 cases of healthy individuals)
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in ctDNA gene and tumor-specific proteins expression | First day in hospital
  Collect 15ml of peripheral blood from subjects, extract ctDNA, and detect mutations in 18 genes (AKT1, APC, BRAF, CDKN2A, CTNNB1, EGFR, FBXW7, FGFR2, GNAS, HRAS, KRAS, NRAS, PIK3CA, PPP2R1A, PTEN, TP53, TOP2A, RNF43) and the expression levels of 9 tumor-specific proteins (CA-125, CA 19-9, CEA, HGF, IL-6, OPN, Prolactin, AFP, HE4) using the FireflyTM method based on amplicon library deep sequencing. Determine the performance indicators including sensitivity, specificity, and accuracy of the existing AccuScreen system and diagnostic model for early screening of gastric cancer. By conducting tests on 10 samples, explore the genomic fragments of gastric cancer, establish targets for ctDNA fragmentomics (fragment length, cleavage sites, end preferences, etc.), and analysis algorithms for gastric cancer fragmentomics, to further evaluate the feasibility of enhancing sensitivity and specificity for early gastric cancer screening through ctDNA fragmentomics detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
This study does not involve clinical trials of drugs; it is solely designed to ensure the confidentiality of patient information. For participant information (such as names and ages), a coding system will be used instead of real names. After enrollment, each case will be assigned an enrollment number. Throughout the entire study, only the main researchers within the research team will have access to participants' real personal data (names, ages) in the electronic database. Distribution and sharing are prohibited. During the publication of articles, the main researchers within the research team will replace participant privacy information (names) with sample codes to achieve de-identification. Furthermore, the protection of participants' personal information will be maintained throughout the study, and any dissemination or leakage is strictly prohibited.